CLINICAL TRIAL: NCT03458338
Title: CKD Prevalence and the Role of Cardiovascular Risk Factors and Infectious Diseases in a Region of Sub-Saharan Africa
Brief Title: Prevalence of Chronic Kidney Disease (CKD) and Risk Factors in Sub-Saharan Africa
Acronym: RenalOne
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss Tropical & Public Health Institute (Other); Ifakara Health Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RenalOne
Record Dates: First submitted 2018-03-01; First posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Chronic Kidney Diseases; Diabetes Mellitus; Hypertension; Tuberculosis; Schistosomiasis; HIV Infections
Keywords: chronic kidney disease; communicable disease; sub-Saharan Africa; Tanzania; neglected disease; prevalence; double burden
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Hypertension; Tuberculosis; Schistosomiasis; HIV Infections; Communicable Diseases; Neglected Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: estimated glomerular filtration rate and albuminuria — chronic kidney disease according to KDIGO

SUMMARY:
Prospective cross-sectional study at the outpatient clinic (OPC) of the Bagamoyo District Hospital (BDH) in Tanzania. Assessment of basic epidemiological data (Point prevalence and risk factors) on CKD with simple clinical, laboratory tests and the patients history. After informed consent blood samples are taken for complete blood count, serum creatinine, HbA1c, HIV-Screening, and urine samples for dipstick, urine sediment, and albumin-creatinine ratio. Further, office blood pressure, weight and height are taken. Further, patients history are asked by a questionnaire (i.e.history of infectious and cardiovascular diseases and basic demographic data: i.e. sex, age).

CKD is defined as the presence of either impaired kidney function and/or albuminuria based on a one-time measurement.

Primary outcome of the study are prevalence rates of CKD and the impact of non-communicable and communicable disorders on CKD.

DETAILED DESCRIPTION:
Study population and Setting:

Single centre cross-sectional study at the outpatient clinic (OPC) of the Bagamoyo District Hospital (BDH) in Tanzania. The BDH is located in Bagamoyo township on the coast of the Indian Ocean and provides care for a semi-rural population. After informed consent, all patients ≥ 18 years, irrespective of the reason of consultation, are included. Pregnant women and patients who are not able or willing to provide an informed signed consent are excluded.

Measurements and procedures:

All data are collected in a case report form, translated from English to Swahili. In all participants body weight and height, blood pressure, heart rate and temperature are recorded. After informed consent, a blood sample is taken for complete blood count and serum creatinine. Complete blood count is performed by a Sysmex Xs 800i analyser. Serum creatinine is measured using Creatinine Jaffe Gen2 reagent on a Cobas Integra 400 plus analyser. HbA1c is measured from capillary blood by using a bed-side DCA 2000+ Analyzer (Siemens Healthcare Diagnostics). After informed consent, HIV-screening is done with an immunochromatographic test for antibodies to HIV-1 and HIV-2 (test kits: Uni-Gold TM HIV, Trinity Biotech, Ireland; Determine® HIV-1/2, Inverness Medical Japan, Japan; SD BIOLINE HIV-1/2 3.0, SD Standard Diagnostics, Korea).

All participants are instructed to void a clean-urine specimen. Urine samples are prepared for microscopic analysis. Albumin-to- creatinine ratio (ACR) is measured using a DCA 2000+ analyser (Siemens Healthcare Diagnostics). CKD is defined as the presence of either impaired kidney function and/or albuminuria based on a one-time measurement. When one-time measurements are used, prevalence of reduced glomerular filtration rate (GFR) and albuminuria might be overestimated due to physiological variation and temporarily elevated values after physical activity and during acute illness or dehydration. Nevertheless, one-time measurements have been used for screening and epidemiologic purposes, as longitudinal documentation is not usually available in epidemiological studies. Kidney function is assessed by eGFR using the CKD-EPI formula. CKD is defined as an eGFR of <60 ml/min/1.73m2 and/or an ACR of ≥30mg/g (≥3 mg/mmol) and categorized according to Kidney Disease: Improving Global Outcomes (KDIGO) stages. Office BP is assessed by a single measurement using a manual sphygmomanometer in a sitting position after 5 minutes at rest. Systolic and diastolic BP is classified as normal (<120/<80 mmHg), pre-hypertensive (120-139/80-89 mmHg), hypertensive stage 1 (140-159/90-99 mmHg) or hypertensive stage 2 (≥160/≥100 mmHg) in analogy to the cut-off values of the JNC 7 report. Anaemia is defined as Hb <13.0 g/dl in male and <12.0 g/dl in female patients. Diabetes mellitus is defined as a history of diabetes, the use of antidiabetic medication or a HbA1c of ≥ 6.5%.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years

Exclusion Criteria:

* pregnant
* not able or willing to provide an informed signed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Single centre cross-sectional study at the outpatient clinic (OPC) of the Bagamoyo District Hospital (BDH) in Tanzania. The BDH is located in Bagamoyo township on the coast of the Indian Ocean and provides care for a semi-rural population. After informed consent, all patients ≥ 18 years, irrespective of the reason of consultation, were included. Pregnant women and patients who were not able or willing to provide an informed signed consent were excluded.
Sampling Method: Probability Sample
Enrollment: 1006 (Actual)
Dates: Start 2010-12-08 (Actual); Primary Completion 2011-05-30 (Actual); Study Completion 2011-05-30 (Actual)

PRIMARY OUTCOMES:
Point prevalence of chronic kidney disease measured by lab values | once measured at baseline, point prevalence
  Measured by serum-creatinine, albuminuria and calculation of estimated glomerular filtration rate (eGFR: serum-creatinine, age, weight, sex)

SECONDARY OUTCOMES:
Risk factors for chronic kidney disease measured by lab values and questionnaire | once measured at baseline
  measurement of HbA1c, haemoglobin, body mass index, sex, age, blood pressure, HIV screening; Questionnaire: patient history of tuberculosis, schistosomiasis, urinary tract infection, known HIV status

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mayr, MD, Principal Investigator — University Hospital Basel, Basel
Locations (1):
- Universitätsspital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hodel NC, Hamad A, Reither K, Mwangoka G, Kasella I, Praehauser C, Abdulla S, Hatz CFR, Mayr M. Assessment of diabetes and prediabetes prevalence and predictors by HbA1c in a population from sub-Saharan Africa with a high proportion of anemia: a prospective cross-sectional study. BMJ Open Diabetes Res Care. 2020 May;8(1):e000939. doi: 10.1136/bmjdrc-2019-000939. PMID 32439737